CLINICAL TRIAL: NCT04551820
Title: SPARC: Study of Peri-operative and Acute Outcomes After Robotic-assisted Cholecystectomy
Brief Title: Study of Peri-operative and Acute Outcomes After Robotic-assisted Cholecystectomy
Acronym: SPARC
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-AHC-2020
Record Dates: First submitted 2020-08-05; First posted 2020-09-16 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Cholecystectomy
MeSH Terms: interventions — After-Hours Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Regular Hours: These subjects have undergone a cholecystectomy during regular hours at the Institution.
  Interventions: Procedure: Regular Hours; Device: Robotic-assisted Cholecystectomy
- After Hours: These subjects have undergone a cholecystectomy during after hours at the Institution.
  Interventions: Procedure: After Hours; Device: Robotic-assisted Cholecystectomy

INTERVENTIONS:
Procedure: Regular Hours — The regular hours cohort includes cholecystectomies performed during the day shift at the Institution during Monday through Friday, not inclusive of national holidays.
  Groups: Regular Hours
Procedure: After Hours — The after hours cohort includes cholecystectomies performed outside of the day shift at the Institution during Monday through Friday, on the weekend, or during a national holiday.
  Groups: After Hours
Device: Robotic-assisted Cholecystectomy — With the patient under general anesthesia, several small incisions are made in the abdomen. Ports are placed, the abdomen is insufflated, and the da Vinci Robotic Surgical System (Intuitive) is docked to the patient and used to complete the cholecystectomy according to the surgeon's standard of care.

SUMMARY:
A multi-center retrospective chart review of short-term outcomes associated with robotic-assisted cholecystectomies performed during regular hours and after-hours.

DETAILED DESCRIPTION:
The study is a retrospective multi-center chart review study of short-term patient outcomes through 30 days after robotic-assisted cholecystectomies performed during regular hours and after-hours. The primary outcomes include the rate of conversion to open, rate of intra-operative adverse events, the rate of post-operative adverse events relating to the cholecystectomy within 30 days, and re-admissions and re-operations relating to the cholecystectomy within 30 days. In addition, operative time, the rate of use of intra-operative imaging, and the hospital length of stay will be collected as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subject between 18 and 80 years of age at the time of surgery.
* Subject underwent a robotic-assisted cholecystectomy during the study time period.

Exclusion Criteria:

* Cholecystectomy was performed as a secondary procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent a robotic-assisted cholecystectomy procedure and meet all eligibility criteria will be considered for enrollment.
Sampling Method: Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Conversion to open | Intra-operative
  The rate of conversion of the cholecystectomy to open, defined as robotic-assisted surgery converted to an open approach.
Number of adverse events | Intra-operative through the 30 day follow-up period
  Intra-operative or post-operative adverse events related to the cholecystectomy
Re-admissions | After discharge from the hospital post-procedure through the 30 day follow-up period
  Re-admissions to the hospital related to the cholecystectomy through the 30 day follow-up period
Re-operations | After the procedure but prior to discharge, through the 30 day follow-up period
  Re-operations related to the cholecystectomy through the 30 day follow-up period

SECONDARY OUTCOMES:
Operative time | Intra-operative
  Operative time, defined as first incision to closure of the incision
Use of intra-operative imaging | Intra-operative
  The rate of use of intra-operative imaging, including indocyanine green fluorescent imaging and cholangiography
Length of Hospital Stay (LOS) | From admission to discharge, up to approximately one week
  How long the patient was admitted to the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- St. David's Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choudhry V, Patel YK, McIntosh BB, Badrudduja M, Jandali M, Vijan S, Brown K. Retrospective multi-center study of robotic-assisted cholecystectomy: after-hours surgery and business-hours surgery outcomes. J Robot Surg. 2024 Jan 20;18(1):48. doi: 10.1007/s11701-023-01765-x. PMID 38244145